CLINICAL TRIAL: NCT06461117
Title: Effect of Beetroot Juice on Anaerobic Performance and Fatigue in Adolescent Male Swimmers
Brief Title: Beetroot Juice: Anaerobic Performance and Fatigue in Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hande Seven Avuk, Head of Nutrition and Dietetic Department, Clinical Assistant Professor, Istanbul Bilgi University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: BEETPERFAS
Record Dates: First submitted 2024-06-07; First posted 2024-06-14 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Nutrition, Healthy
Keywords: sports nutrition; beetroot; nitric oxide; swimming

STUDY DESIGN:
Intervention Model Description: This study designed as a single-blind intervention study.
Who Masked: Participant
Masking Description: Beetroot juice or a placebo drink with the same organoleptic properties was given to the swimmers participating in the study. Participants did not know whether the drink they drank was placebo or beetroot juice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Intervention (No Intervention): In order to determine their standard performance in the first stage before the intervention, the swimmers were subjected to the 8x100 m freestyle maximum effort swimming test at 07:00 on Saturday morning without drinking any beverages. The sets were performed in 2 minutes, and the performance times for each 100-meter run were recorded with a stopwatch. At the end of the 8x100 meter test, the blood lactate values of the swimmers were measured 1 minute later with the Lactate Pro 2 analyzer. Additionally, the Borg Fatigue scale was administered to each swimmer after lactate measurement to measure fatigue levels. After the end of the test, placebo drinks were distributed to the swimmers for the second phase.
  No information was given about whether the drinks given to the swimmers were beet juice or placebo. The swimmers participating in the study were doing double training three days a week and single training on the other days except Sunday.
- Placebo Intervention (Placebo Comparator): In the second stage of the research, swimmers were subjected to the 8x100 m freestyle maximum effort swimming test on the same day and time of the week after consuming a placebo drink. The swimmers' blood lactate values and fatigue scale were reapplied using the same procedure. After the analysis of the results of the placebo intervention, beetroot juice drinks were distributed to the swimmers to be used in the third stage. Swimmers were asked to consume 2x250 ml of beet juice on weekdays and 1x250 ml on Saturdays before the performance test. Swimmers consumed beetroot juice 2.5 hours before training on double training days. On single training days during the week, the patient was asked to consume 2x250 ml of beetroot juice at similar times to other days.
  Interventions: Other: Plesabo Drink
- Beetroot Juice Intervention (Active Comparator): In the third and final stage of the study, the 8x100 meter freestyle maximum effort performance test, blood lactate test, and Borg scale were repeated to make final evaluations of beet juice consumption on the same day and time, and the study was concluded.
  Interventions: Other: Beetroot Juice

INTERVENTIONS:
Other: Beetroot Juice — Beetroot juice (8 mmol NO3-) consumption before training at 6 days
  Arms: Beetroot Juice Intervention
Other: Plesabo Drink — Plesabo drink (0,6 mmol NO3-) consumption before training at 6 days
  Arms: Placebo Intervention

SUMMARY:
The effects of beet juice supplementation on different types of physical performance have been examined in many studies. However, although the number of studies, including the effect of beet juice on physical performance, measuring blood lactate and fatigue levels in swimmers, is limited, most studies focused on acute intake. This study investigated the effects of beetroot juice on anaerobic performance, fatigue, and blood lactate in adolescent male swimmers.Swimmers underwent a single-blind intervention, consuming either a 2x250 ml placebo (0.6 mmol NO3- ) or beetroot juice (8 mmol NO3-) (rich in nitrate, NO3-) for six days. Performance was measured through an 8x100-meter maximal effort swim, with blood lactate and perceived fatigue assessed before and after.

DETAILED DESCRIPTION:
This study, designed as a single-blind intervention study, was conducted in October-November 2023 with adolescent swimmers. . In determining the sample, effect size d (effect size): 1.6975 and standard deviation was taken as 4.12, and the minimum number of samples determined for Power: 0.95 and α: 0.05 in the G*Power 3.1.9 computer program was determined as seven adolescents. Adolescent swimmers with a medical condition diagnosed by a physician, following a special diet, and using regular medication were excluded from the study. Anthropometric measurements (body weight, height, body composition, skin fold measurements), freestyle time trial (TT) swimming performance test, blood lactate measurement and the Borg fatigue scale were taken.

Anthropometric Measurements Body Weight, Height, and Body Composition: The heights of the swimmers were measured with the SECA 213 brand portable stadiometer, with the feet side by side and the head on the Frankfurt plane. Body weight and composition were measured in the morning on an empty stomach, with light clothing, without shoes or socks, using a 0.1 kg sensitive TANITA MC-780 Black professional body composition device.

Skinfold Thickness Measurements: Swimmers' skinfold thicknesses were taken from the triceps, biceps, subscapular, supraspinal, abdomen, thigh, calf, chest, and midaxillary regions using Holstein brand calipers. Measurements were madein accordance with the ISAK protocol (Norton, 2018). The body fat ratio was calculated with the Foulkner (1968) equation, which was developed to calculate the body fat ratio from skinfold thickness measurements on the face.

Freestyle Time Trial (TT) Swimming Performance Test The swimmers' 8x100 m maximum effort swimming performance times were recorded with the help of a Seiko S141 300 memory stopwatch brand stopwatch with 1/100 second precision. A polar watch was attached to the swimmers' right arms, and measurements were taken every 100 m. The start of the performance was made from the sprint stone with the command (take your mark) followed by an electronic beep. 100 m freestyle swimming performance was performed by swimmers with maximum performance.

Blood Lactate Measurement: The blood lactate measurement was completed after the 8x100 m maximum effort swimming performance; blood samples taken from the finger within 10 seconds were analyzed using the Lactate Pro 2 analyzer. Lactate values were recorded in mmol/l.

Borg Fatigue Scale: The level of fatigue perceived by swimmers during the performance was recorded using the "Borg Fatigue Scale." The swimmers were asked to use this scale verbally at the end of each 8x00 meter test, and they were asked to evaluate it between 0 and 10. As the score from the scale increases, the level of perceived fatigue increases (Borg, 1982).

Study Plan:Informed consent forms were obtained after informing the adolescent male swimmers and their parents about the study. Throughout the study, they were instructed to avoid nitrate-rich foods (e.g., beets, celery, spinach). Additionally, they were asked not to use antibacterial mouthwash and chewing gum, which have been shown to kill bacteria in the mouth and impair NO2- bioavailability during the study period (Govoni et al., 2008). In addition, swimmers were asked to stay away from alcohol and tobacco products and maintain their routine eating habits by being able to eat whatever they wanted throughout the study. It was reported that they should avoid consuming caffeine 24 hours before performance tests and consuming anything other than water 3 hours before the test. In addition, swimmers avoided brushing their teeth 24 hours before consumption of sugar, stimulants (e.g., caffeine), or alcohol, using mouthwash, chewing gum, which may alter the oral microbiota and interfere with NO3- reduction (López-Samanes et al., 2020).

This study was conducted in 3 stages to determine the effect of beetroot juice on anaerobic performance and fatigue in adolescent male swimmers.

Pre-Intervention: In order to determine their standard performance in the first stage before the intervention, the swimmers were subjected to the 8x100 m freestyle maximum effort swimming test at 07:00 on Saturday morning without drinking any beverages. The sets were performed in 2 minutes, and the performance times for each 100-meter run were recorded with a stopwatch. At the end of the 8x100 meter test, the blood lactate values of the swimmers were measured 1 minute later with the Lactate Pro 2 analyzer. Additionally, the Borg Fatigue scale was administered to each swimmer after lactate measurement to measure fatigue levels. After the end of the test, placebo drinks were distributed to the swimmers for the second phase.

No information was given about whether the drinks given to the swimmers were beet juice or placebo. The swimmers participating in the study were doing double training three days a week and single training on the other days except Sunday.

Placebo Intervention: In the second stage of the research, swimmers were subjected to the 8x100 m freestyle maximum effort swimming test on the same day and time of the week after consuming a placebo drink. The swimmers' blood lactate values and fatigue scale were reapplied using the same procedure. After the analysis of the results of the placebo intervention, beetroot juice drinks were distributed to the swimmers to be used in the third stage. Swimmers were asked to consume 2x250 ml of beet juice on weekdays and 1x250 ml on Saturdays before the performance test. Swimmers consumed beetroot juice 2.5 hours before training on double training days. On single training days during the week, the patient was asked to consume 2x250 ml of beetroot juice at similar times to other days.

Beetroot Juice Intervention: In the third and final stage of the study, the 8x100 meter freestyle maximum effort performance test, blood lactate test, and Borg scale were repeated to make final evaluations of beet juice consumption on the same day and time, and the study was concluded.

Statistical Analysis: While evaluating the findings obtained in the study, the IBM SPSS Statistics 22 program was used for statistical analysis. The compliance of the parameters with normal distribution was evaluated using the Shapiro-Wilks test. While evaluating the study data, in addition to descriptive statistical methods (minimum, maximum, mean, standard deviation, median, frequency), the Repeated Measures Analysis of Variance test was used for intra-group comparisons of customarily distributed parameters in the comparison of quantitative data, and the Bonferroni test was used as a post hoc test. Friedman Test and Wilcoxon sign test were used as post hoc tests for intragroup comparisons of parameters that did not show normal distribution. Pearson correlation analysis was used to examine the relationships between parameters that conform to normal distribution, and Spearman's rho correlation analysis was used to examine the relationships between parameters that do not comply with normal distribution. Significance was evaluated at p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 ages of adolescent swimmers
* Becoming a licensed swimmer in a sports club

Exclusion Criteria:

* Adolescent swimmers with a medical condition diagnosed by a physician, following a special diet, and using regular medication

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Freestyle Time Trial (TT) Swimming Performance Test | Swimmers' 8x100 m maximum effort swimming performance times were measured and recorded for 3 weeks, before the intervention, on Saturday after consuming placebo drink and beet juice, under similar conditions.
  Performance Test
Blood Lactate Measurement | Blood lactate measurement was measured and recorded before the intervention, after consuming placebo drink and beetroot juice, and after completing the 8x100 m maximum effort swimming performance, under similar conditions, for 3 weeks.
  Blood Lactate Lactate
Borg Fatigue Scale | Swimmers' fatigue was measured for 3 weeks using a Borg Fatigue Scale after performance tests. Minimum and maximum score is 0-10. Higher scores indicate greater fatigue.
  Fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norton KI. Standards for anthropometry assessment. In Kinanthropometry and exercise physiology. 2018; 68-137. Routledge.
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Faulkner JA. Physiology of swimming. Res Q. 1966 Mar;37(1):41-54. No abstract available. PMID 5217133
- [Background] Govoni M, Jansson EA, Weitzberg E, Lundberg JO. The increase in plasma nitrite after a dietary nitrate load is markedly attenuated by an antibacterial mouthwash. Nitric Oxide. 2008 Dec;19(4):333-7. doi: 10.1016/j.niox.2008.08.003. Epub 2008 Aug 30. PMID 18793740
- [Background] Lopez-Samanes A, Gomez Parra A, Moreno-Perez V, Courel-Ibanez J. Does Acute Beetroot Juice Supplementation Improve Neuromuscular Performance and Match Activity in Young Basketball Players? A Randomized, Placebo-Controlled Study. Nutrients. 2020 Jan 9;12(1):188. doi: 10.3390/nu12010188. PMID 31936621